CLINICAL TRIAL: NCT01870713
Title: Serum Proteomics Research in Bypassing Surgery to Treat Type 2 Diabetes in China
Brief Title: Proteomics Study of Gastric Bypass Surgery to Treat Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: No. 150 Central Hospital of the Chinese People Liberation Army (Other Government)
Responsible Party: Sponsor
Other Study IDs: 150CTSX001
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes
Keywords: gastric bypass surgery; proteomics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — whole blood, serum, urine

GROUPS / COHORTS (2):
- type 2 diabetes patients with gastric bypass surgery.: Participants who have type 2 diabetes and with decreased glucose after gastric bypass surgery.
- Weight matched non-operated controls: Participants who are overweight to moderately obese, and have no personal of family history of Type 1, Type 2, or Gestational Diabetes.

SUMMARY:
The purpose of this study is to reveal the key proteins involved in gastric bypassing surgery which may effect the decreased glucose in type 2 diabetes patietns, and evaluate standard remission rate as well as cost-benefit of gastric bypassing surgery for type 2 diabetes mellitus patients in China.

DETAILED DESCRIPTION:
Diabetes Mellitus is a major global problem which responsibles for 4.6 million deaths each year without effective therapy methods. Recently，researchers showed that type 2 diabetes mellitus can be partly reversed by gastric bypassing surgery. However, surgeons are still not clear how to chose the proper diabetes patients for surgery as the mechanism is still not clear, and the remission rate of diabetes mellitus is not the same among different surgical procedures.

This study will enroll type 2 diabetes mellitus patients follwing Roux-en-Y gastric bypassing surgery and obese persons without type 2 diabetes surgery. The defferent expressions of serum proteins of obese persons without type 2 diabetes and type 2 diabetes patients following gastric bypassing surgery after 10 days or 3 months were detected by serum proteomics. Blood samples and urine will be taken prior to surgery, 10 days after surgery and 3 months after surgery. The long term prognosis of diabetes mellitus for 1 years and the remission rate of diabetes of patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as type 2 diabetes are planning to have Roux-en-Y gastric bypass
* age:18-65yr
* HbAlc>8%

Exclusion Criteria:

* diabetes (applies for control patients)
* chronic inflammatory disease
* malignant disease
* pregnancy
* prior gastric, duodenal, proximal jejunal surgery or pancreas resection
* current use of thiazolidinediones
* treatment with incretin mimetics or DPP IV inhibitors in the prior 3 months
* HbAlc<8%
* any condition felt by the investigator to interfere with ability to complete the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients are recruited from No. 150 Central Hospital of PLA
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
different proteins detected between obese persons, type 2 diabetes patients prior to surgery, 10 days after surgery and 3 months after surgery. | base line to 3 months

SECONDARY OUTCOMES:
evaluating the change in glucose between the baseline evaluation and the follow-up evaluation. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- No. 150 Central hospital of Chinese People's Liberation Army, Luoyang, Henan, China